CLINICAL TRIAL: NCT05677282
Title: A Randomized Controlled Trial Evaluating Single-dose Rifaximin Versus Azithromycin With Loperamide Adjunct for Treatment of Acute Watery Diarrhea
Brief Title: Single Dose Antibiotic Treatment of Acute Watery Diarrhea, Rifaximin Versus Azithromycin, With Loperamide Adjunct
Acronym: TrEAT_TD2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Infectious Diseases Clinical Research Program (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDCRP-115
Record Dates: First submitted 2022-11-04; First posted 2023-01-10 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diarrhoea;Acute; Diarrhea Travelers
MeSH Terms: interventions — Rifaximin; Azithromycin; Loperamide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, active-controlled, treatment trial of Travelers Diarrhea (TD) in an outpatient setting enrolling deployed United States (US) service members assigned to Joint Task Force (JTF)-Bravo, Soto Cano Air Base, Honduras and Camp Lemonnier, Djibouti (CLDJ) and United Kingdom (UK) military personnel to British Army Training Unit, Kenya (BATUK) who present for medical care with acute TD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rifaximin with loperamide (Experimental)
  Interventions: Drug: Rifaximin 550 MG; Drug: Loperamide
- Azithromycin mg with loperamide (Active Comparator)
  Interventions: Drug: Azithromycin 500 MG; Drug: Loperamide

INTERVENTIONS:
Drug: Rifaximin 550 MG — Rifaximin 550 mg as a single dose administered orally.
  Arms: Rifaximin with loperamide
Drug: Azithromycin 500 MG — Azithromycin 500 mg as a single dose administered orally.
  Arms: Azithromycin mg with loperamide
Drug: Loperamide — 4 mg loperamide administered orally with study antibiotic (rifaximin or azithromycin). Additional loperamide to use as needed, but not to exceed 16 mg/day for 2 days as per licensed use (one 2 mg capsule after each looses stool).

SUMMARY:
The purpose of this study is to compare a single dose of rifaximin with loperamide to the current standard approach of single dose azithromycin with loperamide for the treatment of acute watery traveler's diarrhea (TD).

The study requires 1) taking a single dose antibiotic plus loperamide to treat TD, 2) providing blood and stool samples at different time points to evaluate infection and immune responses, 3) completing a daily symptom diary following treatment, 4) being seen by the study doctor to monitor illness and recovery, and 5) completing a brief electronic questionnaire at 3 months.

Participants will be randomly assigned to one of the two treatment groups. The two groups are 1) rifaximin 550 mg as a single dose with loperamide 4 mg initially followed by 2 mg after each unformed stool or 2) azithromycin 500 mg as a single dose with loperamide 4 mg initially followed by 2 mg after each unformed stool. Both groups will take the antibiotic dose and 4 mg of loperamide.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty military, 18-60 years old
2. Presence of acute watery diarrhea (3 or more loose/liquid stools in 24 hours or 2 loose/liquid stools in 24 hours and associated symptoms such as nausea, vomiting, abdominal cramps or tenesmus) lasting <96 hours in duration that impacts function in activities and/or performance of primary duties. Refer to recruitment decision tree below.
3. Eligible for ambulatory management. (Note: Ambulatory management in this study means that the patient can be treated on an outpatient basis to include up to 23 hours of medical observation and IV therapies.)
4. Able to comply with follow-up procedures.
5. Will remain in country for at least 7 days or an assurance that follow-up can be arranged elsewhere.

Exclusion Criteria:

1. Allergy to rifamycins, macrolides, or loperamide (not including mild gastrointestinal upset).
2. Antibiotic therapy in the 72 hours prior to presentation (excluding malaria prophylaxis with mefloquine, malarone, chloroquine/proguanil, tafenoquine, or doxycycline).
3. Concomitant medications with known drug-drug interactions with any of the study drugs (includes theophylline, digoxin, warfarin, chloroquine and hydroxychloroquine).
4. Current or history of liver disease or other serious health conditions based on review by study physician.
5. Acute dysentery and/or febrile illness (temperature > 100.4°F [38.1°C]).
6. Presence of symptoms >96 hours prior to initiating treatment.
7. Use of >4 mg loperamide or use of any amount of loperamide for greater than 24 hours prior to enrollment. Prior use of bismuth subsalicylate or other anti-diarrheal, non-antibiotic therapy in the 48 hours prior to enrollment.
8. Positive pregnancy test at presentation (unknown effects with rifaximin). All female participants will be administered a urine pregnancy test prior to enrollment.
9. Previously screened or randomized in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Therapeutic efficacy of single-dose rifaximin (550 mg) with loperamide in treating acute watery diarrhea compared to single-dose azithromycin (500 mg) with loperamide. | Up to 1 week (up to 168 hours)
  Time to last unformed stool (TLUS), in hours, is calculated from the time of antibiotic dose to last unformed (diarrheal) stool (TLUS).

SECONDARY OUTCOMES:
Proportion of participants no longer meeting TD illness criteria at 24 hours | 24 hours
  The clinical efficacy cure rate at 24h is the proportion of participants at the 24h follow up after the initial treatment who met the end point of not meeting TD illness.
Proportion of participants no longer meeting TD illness criteria at 72 hours | 72 hours
  For the clinical efficacy cure rate at 72h is the proportions of participants who met the end point
  1. no report of unformed/diarrheal/loose/liquid stool (LLS) that meet TD illness >24h after initial treatment and
  2. TD-associated symptoms present at 24h were not reported as moderate or greater
Proportion of participants with recurrence of TD illness after previous resolution of TD illness | 7 days
  TD recurrence at 7d follow up if participants meet TD illness and had the previous cure resolution at 24h or 72h
Proportions of serious adverse events (SAE) at 21 days | 21 days
  Proportions of serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Locations (4):
- Camp Lemonnier Djibouti, Djibouti, Djibouti
- JTF-Bravo, Soto Cano AB, Comayagua, Honduras
- British Army Training Site UK, Nanyuki, Kenya
- Fort Magsaysay & Camp Aguinaldo, Santa Rosa, Nueva Ecija, Philippines